CLINICAL TRIAL: NCT06377449
Title: Influence of Ultrasound Examination of the Lungs on the Prognosis and Postoperative Outcomes in Cardiac Surgical Patients
Brief Title: Influence of Lung Ultrasonography on the Prognosis and Postoperative Outcomes in Cardiac Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Filippov Aleksei, MD, PhD, State Cardiovascular Surgeon, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UIL-CSP-18052023
Record Dates: First submitted 2023-11-27; First posted 2024-04-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Heart Disease; Aortic Stenosis, Severe; Aortic Insufficiency; Mitral Stenosis; Mitral Insufficiency; Mitral Stenosis with Insufficiency; Tricuspid Insufficiency; Ascending Aortic Aneurysm
Keywords: Ultrasound examination of the lungs; B-lines; Coronary artery bypass grafting; Heart valve surgery; Cardiopulmonary bypass; On-pump cardiac surgery
MeSH Terms: conditions — Myocardial Ischemia; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Aneurysm, Ascending Aorta

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center study with 2 groups of patients (investigating and control arms)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical management based on results of ultrasound lungs examination (Experimental): Based on the degree/ presence of interstitial pulmonary edema (number of B-lines) and presence of postoperative pleural effusion, identified by regularly performed ultrasound examination of the lungs, medical therapy will be modified in each particular patient to improve clinical status and outcome. Administration of the following drug groups can be made/ doses can be adjusted: Diuretics (furosemide/ Hypothiazide/ spironolactone), Non-steroid antiinflammatory (Ibuprofen), Glucocorticoids.
  Interventions: Diagnostic Test: Ultrasound examination of the lungs
- Medical management based on routine clinical and X-ray diagnostic methods (Active Comparator): Ultrasound examination of the lungs will be performed in all patients in this group, but the attending physician will not be informed about it's results and findings. Any changes in medical therapy/ treatment strategy will be based on standard clinical and X-ray diagnostic methods.
  Interventions: Diagnostic Test: Ultrasound examination of the lungs

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of the lungs — Experimental: Standard ultrasound examination of the lungs based on modified BLUE protocol Active Comparator: Standard ultrasound examination of the lungs based on modified BLUE protocol

SUMMARY:
The goal of this interventional is to assess advantages of the ultrasound examination of the lungs in the early postoperative period in cardiac surgical patients after heart surgeries requiring cardiopulmonary bypass. Evaluation of pulmonary complications and outcomes during mid-term follow-up, as well as comparison of ultrasound examination and traditional roentgenologic methods (X-ray examination and CT of the chest) will be performed. The main question[s] it aims to answer are:

* Is ultrasound examination of the lungs a more specific and sensitive method in identification of early postoperative pulmonary complications after on-pump cardiac surgical procedures, in comparison with traditional X-ray methods.
* Does early identification of interstitial pulmonary edema (based on number of visualised B-lines in the early postoperative period), influences mid-term outcomes in this cohort of patients Participants will undergo ultrasound examination of the lungs on postoperative day 1, 3, 5 and 7 after heart surgery. Based on ultrasound findings and degree of interstitial pulmonary edema, medical (diuretics, anti-inflammatory, e.t.c) therapy will be modified.

Researchers will compare this group of patients with control group, in which ultrasound examination will be performed in the same time frames, but no changes in medical management based on ultrasound findings will be made to see if timely administered medical therapy, based on ultrasound findings, can significantly improve symptoms, hospital lengths of stay and outcomes of this patients.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery with cardiopulmonary bypass (CPB) between 15 December 2023 and 15 December 2024
* signed informed consent for participation in the study

Exclusion Criteria:

* reoperations on the open heart with CPB
* surgical procedures on lungs and lung cancer in the anamnesis
* chronic obstructive pulmonary disease, stage III
* chronic kidney disease, stages 4 and 5
* patients with low Risk Score profile by the Society of Thoracic Surgeons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants with interstitial pulmonary edema at the day of hospital discharge, according to ultrasound lung examination | Ultrasound lung examination every second day of hospital stay; from date of admission until hospital discharge or date of death from any cause, whichever came first, assessed up to 4 weeks
  Participants with more than three B-lines according to ultrasound lung examination (BLUE protocol) at the day of hospital discharge

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Ultrasound lung examination every second day of hospital stay; from date of admission until hospital discharge or date of death from any cause, whichever came first, assessed up to 4 weeks
  Presence of any pulmonary complications (e.g. pleural effusion, pneumothorax, pulmonary edema, atelectasis, pneumonia) during postoperative hospital period will be analyzed
Cumulative dosage of diuretics | Ultrasound lung examination every second day of hospital stay; from date of admission until hospital discharge or date of death from any cause, whichever came first, assessed up to 4 weeks
  Cumulative dosage of administered diuretic drugs will be calculated for each patient in both groups
Number of nights at home after hospital discharge | Ultrasound lung examination every second day of hospital stay; from date of admission until hospital discharge or date of death from any cause, whichever came first, assessed up to 4 weeks
  During 30 days after hospital discharge, the number of nights at home without any additional medical aid due to pulmonary complications, will be found for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Clinic, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not planned to be shared with other parties

REFERENCES:
- [Background] Russell FM, Ehrman RR, Barton A, Sarmiento E, Ottenhoff JE, Nti BK. B-line quantification: comparing learners novice to lung ultrasound assisted by machine artificial intelligence technology to expert review. Ultrasound J. 2021 Jun 30;13(1):33. doi: 10.1186/s13089-021-00234-6. PMID 34191132
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718